CLINICAL TRIAL: NCT03073889
Title: A Comparison Between Scalp Nerve Block and Scalp Infiltration on the Circulatory and Stress Response for Aneurysm Clipping Using an Enhanced Recovery After Surgery Programme
Brief Title: A Comparison Between Scalp Nerve Block and Scalp Infiltration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi Yang (Other)
Responsible Party: Sponsor-Investigator, Xi Yang, Principal Investigator, Wuhan University
Organization: Wuhan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016013
Record Dates: First submitted 2017-01-06; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Aneurysm
Keywords: Aneurysm Clipping; Scalp nerve block; Scalp infiltration; Ropivacaine
MeSH Terms: conditions — Aneurysm | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Block (Experimental): Scalp nerve block with 10ml solution of 0.75% ropivacaine before skin incision, n=15
  Interventions: Procedure: Scalp Nerve Block; Drug: Ropivacaine
- Infiltration (Active Comparator): Scalp infiltration with 10ml solution of 0.75% ropivacaine before incision, n=15
  Interventions: Procedure: Scalp infiltration; Drug: Ropivacaine
- Control (No Intervention): the control group has no treatment, n=15

INTERVENTIONS:
Procedure: Scalp Nerve Block — A scalp nerve block involves regional anesthesia to the nerves that innervate the scalp, including the supraorbital and supratrochlear nerves, branches of the ophthalmic branch of the trigeminal nerve; the zygomaticotemporal nerves, terminal branch of division two of the trigeminal nerve; the auriculotemporal nerves, terminal branch of the mandibular division of the trigeminal nerve; the greater and lesser occipital nerves. The scalp block is performed bilaterally with 10 solution of 0.75% ropivacaine.
  Arms: Block
Procedure: Scalp infiltration — Scalp infiltration before incision. Neurosurgeons infiltrate the planned incision by a 22-gauge needle penetrated deeply to the skin at a 45°angle with 10ml solution of 0.75% ropivacaine throughout the entire thickness of the scalp.
  Arms: Infiltration
Drug: Ropivacaine
  Arms: Block; Infiltration

SUMMARY:
Forty ASA I or II patients, scheduled for aneurysm clipping were enrolled in this prospective, randomized, controlled study. Those patients were randomly divided into 3 groups: Group B (Scalp nerve block before skin incision n=15), Group I (Scalp infiltration before incision n=15), respectively with 0.75% of ropivacaine, and Group C (the control group, n=15). Opioids were used to control haemodynamic responses.All patients received the same general anesthesia.

After intubation, in group B, scalp block was performed by blocking the nerves that innervate the scalp, including the supraorbital, supratrochlear, zygomaticotemporal, auriculotemporal, greater occipital and lesser occipital nerves, and skin along the incision was infiltrated with 0.75% ropivacaine (group I, n = 15), respectively. For group C, there is no treatment. All patients received the same general anesthesia. The depth of anaesthesia was adjusted to maintain a BIS of 40-60. Characteristics of patients were recorded. Heart rate (HR) and mean arterial pressure (MAP) were recorded preoperatively, after induction, before skin incision, the moment of incision, after skin incision. Plasma levels of IL-6, IL-10, CRP were measured before surgery, skin incision,after the surgery. Postoperative pain scores (VAS) for 2, 4, 8, 12, 24, 48 hours after recovery of consciousness were also recorded. Postoperative complications ( nausea, vomiting, infection, and other adverse events) were monitored after surgery.

DETAILED DESCRIPTION:
For group B, the scalp block was performed bilaterally with 0.75% ropivacaine by the anesthesiologist. The supraorbital and supratrochlear nerves emerge from the orbit, and a needle was introduced above the eyebrow perpendicular to the skin with ropivacaine and was then gradually withdrawn with simultaneous injection of solutions throughout the entire. The zygomaticotemporal nerve emerge lateral to the orbit, equal to the position of pterion, this nerve was blocked with ropivacaine. The auriculotemporal nerve was blocked bilaterally anterior to the ear at the level of the tragus, the needle was introduced perpendicularly to the skin and infiltration was performed deep to the fascia and superficially as the needle was withdrawn. Care must be taken to avoid destroying superficial temporal artery. The greater, lesser, and third occipital nerves may be blocked using a needle, with infiltration along the superior nuchal line, approximately halfway between the occipital protuberance and the mastoid process.

For group I patients, neurosurgeons infiltrated the planned incision by a needle penetrated deeply to the skin with 0.75% ropivacaine throughout the entire thickness of the scalp.Neither scalp block nor local infiltration was performed in the control group (group C).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I or II
* Glasgow coma score (GSC) of 15

Exclusion criteria:

* ASA physical status of more than II
* A ruptured cerebral aneurysm and subarachnoid haemorrhage
* A history of allergy to opiates or any other drug used in the study
* Impaired renal, hepatic, or pulmonary function
* Allergic reaction to local anesthetics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change of IL-10 in pg/ml | change from baseline IL-10 values at 24 hour hours after surgery
  Change of plasma levels of IL-10

SECONDARY OUTCOMES:
Change of IL-6 in pg/ml | change for baseline IL-6 values at 24 hour hours after surgery
  Change of plasma levels of IL-6
Mean Arterial Pressure in mmHg | baseline, 5 minutes after induction, 2 seconds after skin incision, 2 minutes and 5 minutes after the incision, 2 seconds after skull drilling
Heart Rate in bpm | baseline, 5 minutes after induction, 2 seconds after skin incision, 2 minutes and 5 minutes after the incision, 2 seconds after skull drilling
Postoperative VAS scores | 2, 4, 8, 12, 24, 48 hours after recovery of consciousness

CONTACTS AND LOCATIONS:
Overall Officials: Mian PENG, Study Chair — Zhongnan Hospital
Locations (1):
- Zhongnan hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leslie K, Troedel S. Does anaesthesia care affect the outcome following craniotomy? J Clin Neurosci. 2002 May;9(3):231-6. doi: 10.1054/jocn.2001.0934. No abstract available. PMID 12093125
- [Background] Quiney N, Cooper R, Stoneham M, Walters F. Pain after craniotomy. A time for reappraisal? Br J Neurosurg. 1996 Jun;10(3):295-9. doi: 10.1080/02688699650040179. PMID 8799542
- [Result] Pakulski C, Nowicki R, Badowicz B, Bak P, Mikulski K, Wojnarska B. Effect of scalp infiltration with lidocaine on the circulatory response to craniotomy. Med Sci Monit. 2001 Jul-Aug;7(4):725-8. PMID 11433201
- [Result] Pinosky ML, Fishman RL, Reeves ST, Harvey SC, Patel S, Palesch Y, Dorman BH. The effect of bupivacaine skull block on the hemodynamic response to craniotomy. Anesth Analg. 1996 Dec;83(6):1256-61. doi: 10.1097/00000539-199612000-00022. PMID 8942596
- [Derived] Yang X, Ma J, Li K, Chen L, Dong R, Lu Y, Zhang Z, Peng M. A comparison of effects of scalp nerve block and local anesthetic infiltration on inflammatory response, hemodynamic response, and postoperative pain in patients undergoing craniotomy for cerebral aneurysms: a randomized controlled trial. BMC Anesthesiol. 2019 Jun 1;19(1):91. doi: 10.1186/s12871-019-0760-4. PMID 31153358